CLINICAL TRIAL: NCT06689956
Title: Outcomes of Low-Risk Endometrial Cancer With Isolated Tumor Cells in the Sentinel Lymph Nodes: a Prospective Multicenter Single-Arm Observational Study
Brief Title: Outcomes of Low-Risk Endometrial Cancer With Isolated Tumor Cells in the Sentinel Lymph Nodes: A Prospective, Multicenter, Single-Arm Observational Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-008963; NCI-2024-09016 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-008963 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: FIGO Grade 1 Endometrial Endometrioid Adenocarcinoma; FIGO Grade 2 Endometrial Endometrioid Adenocarcinoma; Stage IA1 Endometrial Cancer FIGO 2023; Stage IA2 Endometrial Cancer FIGO 2023

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue samples will be collected from sentinel lymph nodes (SLN) biopsy and uterine tumor removed during planned surgery that are not needed for clinical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo tissue sample collection and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study evaluates whether isolated tumor cells in the first lymph nodes near the tumor can tell researchers something important about the future of patients with a certain type of endometrial (uterine) cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether the likelihood of disease recurrence differs between a prospective cohort of patients with low-risk endometrial cancer with ITC and an historical cohort with negative SLNs.

OUTLINE: This is an observational study.

Patients undergo tissue sample collection and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Low-risk endometrial cancer, defined as endometrioid, grade 1 or 2, International Federation of Gynecology and Obstetrics (FIGO) 2009 stage IA (FIGO 2023 stages IA1 and IA2), without substantial/extensive LVSI (≥ 5 vessels involved) at final pathology. Patients with focal LVSI (< 5 vessels involved) will be included.

  * Complete surgical staging, including pelvic sentinel lymph node (SLN) biopsy per National Comprehensive Cancer Network (NCCN) guidelines and ultrastaging.
  * Extent of disease in SLN: ITC (defined as tumor cell aggregates ≤ 0.2 mm or < 200 cells)
  * No adjuvant treatment after surgery
  * Research consent provided.

Exclusion Criteria:

* Prior neoadjuvant chemotherapy.

  * Planning to receive adjuvant treatment.
  * Presence of synchronous cancer (excluding non-melanoma skin cancer).
  * Extent of disease in SLN: micrometastasis (> 0.2 to ≤ 2.0 mm) or macrometastasis (> 2.0 mm).
  * Presence of substantial/extensive LVSI (≥ 5 vessels involved) at final pathology.
  * Prior invasive cancer diagnosis within 5 years of study entry (excluding non-melanoma skin cancer).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with low-risk endometrial cancer.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | Up to 5 years
  RFS is defined as the length of time after primary treatment that the patient survives without any signs or symptoms of that cancer. (Recurrence may be vaginal, hematogenous, lymphatic, or peritoneal.) RFS will be measured from the date of surgery to the date of recurrence, death, or last disease evaluation.

SECONDARY OUTCOMES:
Non-vaginal RFS | Up to 5 years
  Non-vaginal RFS is defined as the interval from the date of surgery to the date of the first of the following events: non-vaginal recurrence or death due to any cause.
Overall Survival (OS) | Up to 5 years
  Overall survival is defined as the time from surgery to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen E. Glaser, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (20):
- United States (3):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Houston Methodist Hospital, Houston, Texas
- Medical University of Vienna, Vienna, Austria
- AC Camargo Cancer Center, São Paulo, Brazil
- Canada (2):
  - Sunnybrook Health Sciences, University of Toronto, Toronto, Ontario
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
- Institut Universitaire du Cancer Toulouse Oncopole, Toulouse, France
- University Hospital Essen, Essen, Germany
- Meir Medical Center, Faculty of Medicine - Tel-Aviv University, Kefar Sava, Israel
- Italy (7):
  - Ospedale Michele e Pietro Ferrero, Verduno, CN
  - IRCCS Fondazione San Gerardo dei Tintori, Monza, MB
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan, MI
  - European Institute of Oncology, Milan, MI
  - Policlinico Universitario Fondazione Agostino Gemelli, Roma, RM
  - University of Udine, Udine, UD
  - Istituto Nazionale Tumori, IRCCS, Fondazione G. Pascale, Naples
- Spain (2):
  - Hospital Materno of Las Palmas, Las Palmas
  - Hospital Universitario La Paz, Madrid
- Ospedale Regionale di Lugano, Civico, Lugano, Switzerland

REFERENCES:
- [Derived] De Vitis LA, Bogani G, Raspagliesi F, Arencibia Sanchez O, Navarro B, Multinu F, Zanagnolo V, Baiocchi G, De Brot L, Fanfani F, Capasso I, Piedimonte S, DeGuerke L, Buda A, Mauro J, Alessio M, Filipello F, Beiner M, Kadan Y, Papadia A, Vizzielli G, Restaino S, Grassi T, Landoni F, Bianchi T, Grimm C, Polterauer S, Ricotta G, Martinez A, Buderath P, Kimmig R, Chiantera V, Zand B, Zapardiel I, Hernandez A, Gill S, Covens A, Dagher C, Meschini T, Cucinella G, Schivardi G, Occhiali T, Lembo A, Palmieri E, Shahi M, Fought AJ, McGree ME, Suman VJ, Abu-Rustum NR, Ramirez PT, Mariani A, Glaser GE; Low Volume Metastasis in Endometrial Cancer Consortium. Outcomes of low-risk endometrial cancer with isolated tumor cells in the sentinel lymph nodes: a prospective, multi-center, single-arm, observational study (ENDO-ITC study). Int J Gynecol Cancer. 2025 Aug;35(8):101764. doi: 10.1016/j.ijgc.2025.101764. Epub 2025 Mar 7. PMID 40148176
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials